CLINICAL TRIAL: NCT05002101
Title: The Effect of Daily Zinc Supplementation on Prevention of Diarrhea and Acute Respiratory Infections Among Children Less Than Five Years: A Randomized Controlled Trial
Brief Title: Daily Zinc Supplement Effect on Prevention of Diarrhea and Acute Respiratory Infections in Children Less Than Five Years
Acronym: RCTZ
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Yosra Samir Abd El Ghaffar Souliman, Assistant lecturer of public health - Department of Community, Environmental and Occupational Medicine, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MD180 2018
Record Dates: First submitted 2021-07-26; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Zinc Deficiency; Child Nutrition Disorders
Keywords: zinc; diarrhea; Respiratory Tract Infections; prevention
MeSH Terms: conditions — Child Nutrition Disorders; Diarrhea; Respiratory Tract Infections | interventions — Zinc; Zinc Sulfate

STUDY DESIGN:
Who Masked: Participant
Masking Description: The study was single-blinded, where the children's mothers didn't know either their children are enrolled in the study group or the control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- zinc group (Active Comparator): The children were randomized to receive daily zinc sulphate. The elemental zinc dose was 3 mg/ day to children whose weight is less than 10 kg and 7 mg/ day to children whose weight is 10 kg or more.
  Interventions: Dietary Supplement: zinc
- placebo group (Placebo Comparator): The placebo was non-nutritious and vitamin-free, designed to be identical to the zinc syrup in colour, odour, consistency and taste. Zinc and placebo syrups were packaged in similar bottles.
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: zinc — The zinc syrup was prepared with a concentration of 7 mg zinc in each 5 ml solution. Accordingly, children with weight more than 10 kg were asked to take 5 ml syrup daily, while children with weight less than 10 kg were asked to take 2.5 ml daily.
  Other Names: zinc sulphate
  Arms: zinc group
Drug: Placebo — Children with weight more than 10 kg were asked to take 5 ml syrup daily, while children with weight less than 10 kg were asked to take 2.5 ml daily.
  Other Names: inactive substance
  Arms: placebo group

SUMMARY:
Zinc deficiency in children is a major problem which leads to compromised immunity and accordingly repeated infections. This study aims to investigate the effect of supplementing zinc to decrease the incidence of diarrhea and respiratory illness in children between 6 months and 5 years in Paediatric Outpatient Clinic in Ain Shams University Hospital.

DETAILED DESCRIPTION:
Zinc is a trace element that plays essential roles in protein and lipid metabolism, cell growth and differentiation, and the immune system; either cellular or humoral immunity. There is no specialized zinc storage system in the body, accordingly, a daily intake of zinc is required to maintain a steady state. Zinc deficiency can cause compromised immune function, accordingly this can lead to infections and growth defects among young children According to literature review search, there is lack of studies on the preventive effect of zinc supplementation on Egyptian children less than five years old; the age group which is known by the suboptimal nutritional status and the high prevalence of infection. Accordingly, the present study is aiming to evaluate the impact of 4 months of daily zinc supplementation on the incidence of diarrhea and respiratory illness and to detect the frequency of daily dietary intake of zinc-rich food children between 6 months and 5 years in Paediatric Outpatient Clinic in Ain Shams University Hospital.

Objectives:

1. To evaluate the impact of 4 months of daily zinc supplementation on:

   - the incidence and the severity of diarrheal morbidity.

   - the incidence of acute respiratory infection.
2. To measure the level of serum zinc in children between 6 months and 5 years attending Paediatric Outpatient Clinic in Ain Shams University Hospital.
3. To compare between children who had initially low serum zinc level with those with normal level as regard the reduction in the incidence of diarrhea and respiratory illness.
4. To measure the frequency of daily dietary intake of zinc-rich food in children between 6 months and 5 years attending Paediatric Outpatient Clinic in Ain Shams University Hospital.

   Methodology:

   • Study type: a single blinded, randomized controlled trial.

   • Study setting: Paediatric Outpatient Clinic in Ain Shams University Hospital.
   * Sampling method:

   A convenience sample of children between 6 months and 5 years was recruited from the Paediatric Outpatient Clinic in Ain Shams University Hospital.

   • Study population: Eligible children aged between 6 months and 5 years attending Paediatric Outpatient Clinic in Ain Shams University Hospital was included.

   Randomization and allocation:

   Random assignment of the sampled children to either the study group receiving zinc or the control group receiving placebo was done. The study was single-blinded, where the children's mothers won't know either their children are enrolled in the study group or the control group.

   • Study tool:

   - Baseline questionnaire: Structured interview questionnaire was used at the first meeting with the mother to collect baseline data. The questionnaire includes baseline characteristics, such as child age, child sex, family size, child rank, child feeding practices (breastfeeding), maternal literacy, vaccination history and birth weight.

   Also, the baseline questionnaire assessed the occurrence and duration of diarrhea and respiratory illness in the past month before the start of zinc supplementation. Questions are adopted from the Demographic and Health Survey (DHS) questionnaire (Ministry of Health and Population/Egypt, 2015).

   - Questionnaire for Zinc-Rich Food Intake Pattern:

   The questionnaire, a dietary history recall instrument, was used to elicit and capture information on frequency of daily dietary intake over previous 1 month of two categories of zinc-rich foods namely:
   * Foods of animal origin devoid of zinc antinutritional factor (liver, fish, milk, eggs)
   * Food of vegetable origin including those known to contain a zinc antinutritional factor (cereals, beans)

     - Serum zinc: A blood sample was collected from all included children at the beginning of the study to estimate the baseline serum zinc level. Venous blood samples (about 4 milliliters) were collected in heparinised tubes and transported to the laboratory for centrifugation and serum zinc estimation using atomic absorption spectrophotometer graphites.

     - Intervention: The children were randomized to receive daily zinc sulphate or placebo. The elemental zinc dose was 3 mg/ day to children whose weight is less than 10 kg and 7 mg/ day to children whose weight is 10 kg or more. This dose is more than the recommended dietary allowance for supplementation so as to allow for possible impairment in absorption of ingested zinc among children as a result of consumption of a predominantly phytate-rich cereal-based diet, bacterial overgrowth, and protozoal or parasitic infestations. At the same time the dose won't exceed the upper tolerable level for zinc (World Health Organization and Food and Agriculture Organization of the United Nations, 2005).

   One bottle that contained 150 mL was kept in the child's home and replaced monthly. The placebo was non-nutritious and vitamin-free, designed to be identical to the zinc syrup in colour, odour, and taste.

   - Follow up: Each month, during the child visit to the Paediatric Outpatient Clinic, or through a telephone call, the mother was asked certain questions regarding the occurrence and duration of diarrhea and respiratory illness in the past month. Questions are adopted from the Demographic and Health Survey (DHS) questionnaire (Ministry of Health and Population/Egypt, 2015).

   - Pre- and posttreatment anthropometric parameters (weight and length\ height measurements) were recorded.

   Nutritional status was assessed by measuring weight and height using standard methods and calculating weight for-age and weight-for-height Z scores. Weight was measured to nearest 100 gm using an electronic scale.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy child with good general health

Exclusion Criteria:

* Children with severe malnutrition requiring hospital admission,
* Cases of chronic and metabolic diseases as diabetic children
* Children suffering from any type of cancer or any other debilitating disease.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Change in the baseline cumulative incidence rate of diarrhea at 4 months | after 4 months
  Cumulative incidence rate of diarrhea at the baseline before intervention was compared to the cumulative incidence rate of diarrhea after 4 months of daily zinc supplements administration
Change in the baseline cumulative incidence rate of acute respiratory infections at 4 months | after 4 months
  Cumulative incidence rate of acute respiratory infections at the baseline before intervention was compared to the cumulative incidence rate of acute respiratory infections after 4 months of daily zinc supplements administration.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed E Shouman, Professor, Study Director — Faculty of Medicine, Ain-Shams University
Locations (1):
- Pediatric outpatient clinic in Ain Shams University hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liberato SC, Singh G, Mulholland K. Zinc supplementation in young children: A review of the literature focusing on diarrhoea prevention and treatment. Clin Nutr. 2015 Apr;34(2):181-8. doi: 10.1016/j.clnu.2014.08.002. Epub 2014 Aug 13. PMID 25176404
- [Derived] Abd El-Ghaffar YS, Shouman AE, Hakim SA, El Gendy YGA, Wahdan MMM. Effect of Zinc Supplementation in Children Less Than 5 Years on Diarrhea Attacks: A Randomized Controlled Trial. Glob Pediatr Health. 2022 Jun 17;9:2333794X221099266. doi: 10.1177/2333794X221099266. eCollection 2022. PMID 35747897